CLINICAL TRIAL: NCT05799014
Title: The Effectiveness and Safety of Percutaneous Lung Biopsy Guided by Electromagnetic Navigation Real-time Positioning Technology
Brief Title: The Effectiveness and Safety of Electromagnetic Navigation Real-time Guided Percutaneous Lung Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-NHLHCRF-LX-01-0201-01
Record Dates: First submitted 2023-03-08; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Lung Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional CT-guided percutaneous lung biopsy group (Experimental)
  Interventions: Procedure: CT-guided percutaneous lung biopsy
- Percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology group (Experimental)
  Interventions: Procedure: Percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology

INTERVENTIONS:
Procedure: CT-guided percutaneous lung biopsy — The participants would undergo CT-guided percutaneous lung biopsy.
  Arms: Traditional CT-guided percutaneous lung biopsy group
Procedure: Percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology — The participants would undergo percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology.
  Arms: Percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology group

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic efficacy and safety of percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology in peripheral lung lesions. The main question it aims to answer are: the effectiveness and safety of percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology.

Participants will undergo CT-guided percutaneous lung biopsy or percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Imaging examination showed peripheral lung lesions
* Selected patients need to complete routine preoperative examinations such as blood routine examination, coagulation function, electrocardiogram, chest CT, etc
* There is no contraindication for puncture biopsy
* Good compliance, able to cooperate with research and observation
* Fully informed of the purpose and method of the study, agreed to participate in the study, and signed the informed consent form

Exclusion Criteria:

* Severe cardiopulmonary insufficiency, extreme weakness and intolerance of patients
* The patient is allergic to lidocaine and midazolam
* The site to be biopsied has a high risk of bleeding such as bronchial artery penetration or suspected lung metastasis of renal cancer
* Unstable angina pectoris, congestive heart failure, severe bronchial asthma
* The patient did not agree to participate in the study
* Participation in other studies within three months without withdrawal or termination will affect the observation of this study
* The researcher believes that there is any person who is not suitable for the selection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology for diagnosis of pleural effusion. | 7 days after the lung biopsy
  The diagnosis would be confirmed according to the pathological results or multidisciplinary discussion results (if interstitial lung disease is suspected, the multidisciplinary discussion results shall be recorded).
  The diagnostic efficacy of percutaneous lung biopsy guided by electromagnetic navigation real-time positioning technology will be compared with that of CT-guided percutaneous lung biopsy for diagnosis of pleural effusion.

SECONDARY OUTCOMES:
Operation time | during the operation of lung biopsy
  Timer